CLINICAL TRIAL: NCT04756557
Title: Caries-preventing Effect of a Hydroxyapatite-toothpaste in Adults
Acronym: CA1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: Medical University of Bialystok (Other); Dr. Kurt Wolff GmbH & Co. KG (Industry)
Responsible Party: Principal Investigator, Elzbieta Paszynska, Head of Department of Integrated Dentistry, Principal Investigator, Clinical Associate Professor, Poznan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PoznanUMS
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Dental Caries; Hydroxyapatite; Tooth Decay; Dentin, Carious; Enamel Caries
Keywords: tooth demineralization; cariostatic agent; protective agent; toothpaste
MeSH Terms: conditions — Dental Caries; Tooth Demineralization | interventions — Durapatite

STUDY DESIGN:
Intervention Model Description: Multicenter, double-blind, randomized, active-controlled parallel-group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) The study will be double-blinded (blinded for the study subjects as well as for the investigators). The blind must not be broken throughout the study. Only after study end, study subjects will be informed on the toothpaste received, if requested by the subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tooth Brushing HAP Toothpaste (Experimental): Experimental: Tooth Brushing HAP HAP-Toothpaste Tooth Brushing HAP Prophylactic cleaning of all teeth using a standardized electric tooth brush and a non-fluoridated toothpaste containing microcrystalline hydroxylapatite two x daily over the duration of the study (18 months).
  Procedure: Tooth Brushing HAP
  Interventions: Other: Experimental.
- Tooth Brushing F Toothpaste (Active Comparator): Cleaning teeth using a standardized electric tooth brush and a fluoridated tooth paste containing amino fluoride (1450 ppm F-), (two x daily over the duration of the study (18 months).
  Interventions: Other: Active comparator

INTERVENTIONS:
Other: Experimental. — Tooth Brushing HAP 2x daily repeated cleaning of all teeth 3 min. using a standardized electric tooth brush Electric (powered) toothbrushes (Oral-B; P&G, Schwalbach, Germany), brushing head: medium; will be changed every 2 months and a non-fluoridated tooth paste containing microcrystalline hydroxyapatite . HAP-toothpaste (Karex toothpaste with 10 % hydroxyapatite) If a subject shows multiple carious lesions during the course of the study, the study dentist will decide whether the subject must be excluded from the study. In this case the subject will receive additional intensive caries prophylactic measures (e.g. chlorhexi-dine gel application, dietary counselling, etc.). Caries preventive treatment (removing caries and placing a restoration) by the study centers is offered.
  Other Names: Karex Toothpaste with 10% Hydroxyapatite
  Arms: Tooth Brushing HAP Toothpaste
Other: Active comparator — Tooth Brushing F 2x daily repeated cleaning of all teeth 3min.using a standardized electric tooth brush ((Oral-B; P&G, Schwalbach, Germany) and a fluoridated toothpaste (Karex Base with sodium fluoride 1450 F-), brushing head: medium; will be changed every 2 months If a subject shows multiple carious lesions during the course of the study, the study dentist will decide whether the subject must be excluded from the study. In this case the subject will receive additional intensive caries prophylactic measures (e.g. chlorhexidine gel application, dietary counselling, etc.). Caries preventive treatment (removing caries and placing a restoration) by the study centers is offered.
  Other Names: Karex Base with sodium fluoride 1450 F-
  Arms: Tooth Brushing F Toothpaste

SUMMARY:
Target question is as the following one:

Does the daily use of a fluoride-free, microcrystalline hydroxyap-atite (HAP) - containing test toothpaste have a non-inferior caries preventing effect in the permanent dentition compared to the regular use of a fluoride control toothpaste (1450 ppm F-) with proven caries preventive efficacy (Walsh et al. 2019)? This multicenter, non-inferiority clinical trial, randomized, double-blind, active-controlled design, two-armed study evaluates the hypothesis that the home regular use of a toothpaste containing microcrystalline hydroxylapatite (HAP) (test toothpaste) provides a caries preventive effect in adults aged 18-45 comparable to the caries preventive effect provided by the regular use of a fluoridated tooth paste (1450 ppm -F) (control toothpaste) over observation periods of max. 18 months. Caries development will be assessed according to the clinical criteria of the Decay Missing Filling Surface Index (DMFS).

DETAILED DESCRIPTION:
Caries-preventing effects of hydroxyapatite toothpastes have been shown in vivo [children and adolescents] (Schlagenhauf et al. 2019, Paszynska et al. 2021), in situ (Amaechi et al. 2019), and in vitro (Tschoppe et al. 2011). However, to date, the caries-preventing effect of a hydroxyapatite toothpaste in adults (without orthodontic treatment) has not been investigated in a clinical trial compared to fluoride toothpastes.

The aim of this clinical trial is to assess in cohorts of adults whether 2 x daily tooth brushing at home over an observation period of 18 months with a fluoride-free, microcrystalline hydroxyapatite (HAP) - containing test toothpaste has a non-inferior caries preventing effect in the permanent dentition compared to the regular use of a fluoride control toothpaste (1450 ppm F-) with proven caries preventive efficacy (Walsh et al. 2019). The study is designed as a multicentre, two armed, non-inferiority trial and will be performed by 2 study centres in Poland. Caries development will be assessed by the Decay Missing Filling Surface Index (DMFS).

There are planned 4 visits for all subjects included to the project. Description of the 4 visits is presented below.

Visit 1 (Screening and Baseline): Study day 0, informed consent, screening, collection of baseline data, and study inclusion Subjects potentially suitable for the study will be informed by the investigator about the nature, sig-nificance, and scope of the clinical trial according to the requirements described in the written subject information.

Before study inclusion, the willingness of the subjects to properly follow the study protocol during the complete treatment period of 546 days must be assessed. Only when subjects have given their written informed consent, he/she will be included as study participant.

Subjects have to meet all inclusion criteria and no exclusion criteria. Unsuitable subjects with un-treated caries in need of a restoration can become eligible after restorative therapy.

Once informed consent has been given, an initial examination will take place that covers the follow-ing aspects:

* Screening subjects for study eligibility (inclusion and exclusion criteria)
* Demographic data Assessment of the study parameters has to be done on all teeth in the following sequence
* Plaque control record (PCR)
* Professional tooth cleaning
* DMFS
* DIAGNOcam After the analysis of the plaque control record using a plaque-staining solution (see O' Leary T, Drake R, Naylor, 1972), a professional tooth cleaning will be performed. Thereafter, no fluoride gel/varnish etc. will be applied.

Finally, the study subjects receive an electric toothbrush with 3 brushing heads (replacement of the brushing head every 2 months) and the allocated toothpaste (test or control) by a trained study nurse or dentist not involved in clinical study examinations.

Proper use of the assigned electric toothbrush and the issued toothpaste is also instructed by this study nurse or a dentist not involved in the clinical study examinations.

Visit 2: Study day 182 (± 28 days at most), 1st follow-up examination 182 days after baseline visit the following parameters are reassessed:

* Plaque control record (PCR)
* Caries status (DMFS) as described for the baseline visit. Subsequently a study nurse or a dentist not involved in clinical study examinations will hand out 3 new brushing heads for the electric toothbrush and a new supply of the assigned experimental toothpaste (test or control) for the next 182 days.

Furthermore, the study nurse will subsequently check the efficacy of the oral hygiene efforts of the subjects and if PCR will be > 15%, will train again with the subjects an efficacious brushing tech-nique. Finally, subjects receive a new appointment for visit 3.

Visit 3: Study day 364 (± 28 days at most), 2nd follow-up examination 364 days after baseline visit the following parameters are reassessed:

* Plaque control record (PCR)
* DMFS as described for the baseline visit. Subsequently a study nurse or a dentist not involved in the clinical study examinations will hand out 3 new brushing heads for the electric toothbrush and a new supply of the assigned experimental toothpaste (test or control) for the next 182 days.

Furthermore, the study nurse will subsequently check the efficacy of the oral hygiene efforts of the subjects and if PCR will be > 15%, will train again with the subjects an efficacious brushing tech-nique. Finally, subjects receive a new appointment for visit 4.

Visit 4: Study day 546 (± 28 days at most), final visit 546 days after baseline visit the following assessments are repeated:

* Plaque control record (PCR)
* Professional tooth cleaning
* DMFS
* DIAGNOcam as described for the baseline visit.

Methods of Determining Efficacy and Safety Methods of Determining Efficacy DMFS-index and PCR-scores will be determined by clinical examinations of the oral cavity. In addi-tion, analysis of mineral density using DIAGNOcam will be conducted according to the instructions of the manufacturer.

Assessments of all clinical findings will be performed only by experienced dentists.

DMFS Index Calculation The DMFS Index (Decayed Missed Filled Surfaces) is one of the most common methods in oral epidemiology for assessing dental caries prevalence as well as dental treatment needs among populations.

DMFS Index calculation: There are five surfaces on the posterior teeth: facial, lingual, mesial, distal, and occlusal. There are four surfaces on anterior teeth: facial, lingual, mesial, and distal. The third molars are not counted.

* When a carious lesion or both a carious lesion and a restoration are present, the surface is listed as a D.
* When a tooth has been extracted due to caries, it is listed as an M.
* When a permanent filling is present, or when a filling is defective but not decayed, this surface is counted as an F. Surfaces restored for reasons other than caries are not counted as an F.

The total count is 128 surfaces.

DIAGNOcam (KaVo Dental) DIAGNOcam will be used according to the instructions of the manufacturer. The following classifi-cation will be used (Dent. Med. Probl. 2016, 53, 4, 468-475).

0 = Light transmission unchanged

1. = Shadow visible in enamel
2. = Shadow visible in dentin

Plaque Control Record The Plaque Control Record (O' Leary T, Drake R, Naylor, 1972) is a simple method of recording the presence of the plaque on individual tooth surfaces.

At the study visits a suitable disclosing solution such as Bismarck Brown, Diaplac or similar is painted on tooth surfaces. After the subject has rinsed, the investigator (using an explorer or a tip of a probe) examines each stained surface for soft accumulations at the dentogingival junction.

After all teeth are examined and scored, the index is calculated by dividing the number of plaque containing surfaces by the total number of available surfaces.

Plaque Index Calculation = The number of plaque containing surfaces / The total number of available surfaces

ELIGIBILITY:
Inclusion Criteria:

* provision of written informed consent
* age 18-45 years (both men and women)
* a minimum of 10 healthy molars and premolars (DMFS of these teeth = 0)
* willing to use an electric (powered) toothbrush

Exclusion Criteria:

* Medical Reasons

  * untreated caries [clinical investigation and analysis with DI-AGNOcam] (→ unsuitable subjects with untreated caries in need of a restoration can become eligible after restorative therapy)
  * severe periodontitis at the baseline-visit (pocket depth on at least one tooth ≥ 5.5 mm)
  * orthodontic treatment
  * known hypersensitivity to one of the ingredients of the tooth-pastes to be tested
  * systemic disorders interfering with salivary function or flow
  * regular medication intake interfering with salivary function or flow
* Other Reasons:

  * Participation in any other clinical study within the past 3 months or ongoing
  * lack of intellectual or physical ability to conduct the study properly
  * Any other reason that, in the opinion of the investigator, dis-qualifies the subject from participating in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects showing no increase in overall DMFS-index | 546 days
  Proportion of subjects showing no increase in overall DMFS-index (DMFSVisit 4 - DMFSVisit 1 = 0) during the observation period

SECONDARY OUTCOMES:
roportion of subjects experiencing no change in mineral density | 546 days
  A) Proportion of subjects experiencing no change in mineral density (as analyzed by DIAGNOcam) during the observation period of time
Changes in the coverage of all teeth with bacterial plaque ac-cording to the criteria of the Plaque Control Record | 546 days
  B) Changes in the coverage of all teeth with bacterial plaque ac-cording to the criteria of the Plaque Control Record (PCR; O'Leary et al. 1972)

CONTACTS AND LOCATIONS:
Overall Officials: Elzbieta Paszynska, Prof, Principal Investigator — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No
we do not plan any individual participant data available data to other researchers

REFERENCES:
- [Background] Walsh T, Worthington HV, Glenny AM, Marinho VC, Jeroncic A. Fluoride toothpastes of different concentrations for preventing dental caries. Cochrane Database Syst Rev. 2019 Mar 4;3(3):CD007868. doi: 10.1002/14651858.CD007868.pub3. PMID 30829399
- [Result] Piaggio G, Elbourne DR, Pocock SJ, Evans SJ, Altman DG; CONSORT Group. Reporting of noninferiority and equivalence randomized trials: extension of the CONSORT 2010 statement. JAMA. 2012 Dec 26;308(24):2594-604. doi: 10.1001/jama.2012.87802. PMID 23268518
- [Result] Paszynska E, Pawinska M, Gawriolek M, Kaminska I, Otulakowska-Skrzynska J, Marczuk-Kolada G, Rzatowski S, Sokolowska K, Olszewska A, Schlagenhauf U, May TW, Amaechi BT, Luczaj-Cepowicz E. Impact of a toothpaste with microcrystalline hydroxyapatite on the occurrence of early childhood caries: a 1-year randomized clinical trial. Sci Rep. 2021 Jan 29;11(1):2650. doi: 10.1038/s41598-021-81112-y. PMID 33514787
- [Result] Amaechi BT, AbdulAzees PA, Alshareif DO, Shehata MA, Lima PPCS, Abdollahi A, Kalkhorani PS, Evans V. Comparative efficacy of a hydroxyapatite and a fluoride toothpaste for prevention and remineralization of dental caries in children. BDJ Open. 2019 Dec 9;5:18. doi: 10.1038/s41405-019-0026-8. eCollection 2019. PMID 31839988
- [Result] Hummel R, Akveld NAE, Bruers JJM, van der Sanden WJM, Su N, van der Heijden GJMG. Caries Progression Rates Revisited: A Systematic Review. J Dent Res. 2019 Jul;98(7):746-754. doi: 10.1177/0022034519847953. Epub 2019 May 9. PMID 31070943
- [Result] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- [Result] Poulsen VJ. Caries risk children in the Danish child dental service. Scand J Prim Health Care. 1987 Sep;5(3):169-75. doi: 10.3109/02813438709013999. PMID 3671918
- [Result] Tschoppe P, Zandim DL, Martus P, Kielbassa AM. Enamel and dentine remineralization by nano-hydroxyapatite toothpastes. J Dent. 2011 Jun;39(6):430-7. doi: 10.1016/j.jdent.2011.03.008. Epub 2011 Apr 8. PMID 21504777
- [Derived] Paszynska E, Pawinska M, Enax J, Meyer F, Schulze Zur Wiesche E, May TW, Amaechi BT, Limeback H, Hernik A, Otulakowska-Skrzynska J, Krahel A, Kaminska I, Lapinska-Antonczuk J, Stokowska E, Gawriolek M. Caries-preventing effect of a hydroxyapatite-toothpaste in adults: a 18-month double-blinded randomized clinical trial. Front Public Health. 2023 Jul 18;11:1199728. doi: 10.3389/fpubh.2023.1199728. eCollection 2023. PMID 37533523